CLINICAL TRIAL: NCT05710211
Title: Clonal Architecture of ASXL1-mutated Myelofibrosis
Acronym: CLONEMF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A02497-36
Record Dates: First submitted 2022-12-28; First posted 2023-02-02 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CLONEMF cohort (Experimental)
  Interventions: Biological: Clonal architecture determination

INTERVENTIONS:
Biological: Clonal architecture determination — Biological:
  * Determination of clonal architecture by sorting of circulating CD34 positive cells followed by cell culture and colony genotyping and/or single-cell DNA-sequencing
  * Secondary outcome: transcriptomic study by RNA-sequencing

SUMMARY:
Prospective study to decipher the clonal architecture of ASXL1-mutated primary and secondary myelofibrosis and its impact on prognosis

DETAILED DESCRIPTION:
The clonal architecture of myelofibrosis patients is still little described. Inconsistent results in terms of the prognostic value of some mutations are observed in the literature, in particular concerning ASXL1 mutations. We assume that a better understanding of the clonal architecture of ASXL1-mutated myelofibrosis could help refining the prognostic impact of ASXL1 mutations.

This study aims to evaluate a multicenter cohort of 50 patients. Blood of patients will be collected within 18 months of diagnosis. After 4 years of follow-up of the patient as part of his usual care, data on survival and leukemic transformation will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years),
* Affiliated to the national social security system,
* ASXL1 mutated primary or secondary myelofibrosis,
* Signed the consent to participate in the study,
* Included, or consenting to be included, in the national clinical-biological database of France Intergroupe Syndrome Myéloprolifératifs (FIM).

Exclusion Criteria:

* Patient with another active hematological disease or cancer at the time of diagnosis,
* Person subject to legal protection scheme or incapable of giving consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Identify subgroups of ASXL1-mutated myelofibrosis based on clonal architecture data | 24 months
  The clonal architecture is defined by the number of mutations (numerical), the order of acquisition of the mutations (categorial, pre/post/separated), the mutational branching (categorial, yes/no), the presence of distinct clones (categorial, yes/no) and the transition towards homozygosity of each clone (categorial, yes/no). All parameters of clonal architecture will be analyzed together using a multivariate classification (Factor Analysis for Mixed Data) followed by a clustering which allow us to identify homogeneous cluster of patients.

SECONDARY OUTCOMES:
Description of previously constituted prognostic genomic groups (according to Luque Paz et al. 2021) within identified clusters of clonal architecture | 24 months
  The repartition of patients onto genomic groups will be reported for each clusters of clonal architecture (number and percentage).
Studying the functional characteristics of each subtype of clonal architecture by transcriptomics | 24 months
  Gene Set Enrichment Analysis (GSEA) will be performed for each cluster of clonal architecture
Comparison of male proportion within the subtypes of clonal architecture | 24 months
  Repartition of gender will be compared
Comparison of age at the time of diagnosis within the subtypes of clonal architecture | 24 months
  Age at the time (years) of diagnosis will be compared
Comparison of blood counts within the subtypes of clonal architecture | 24 months
  Blood counts (g/dL or G/L) at the time of diagnosis will be compared
Comparison of LDH levels within the subtypes of clonal architecture | 24 months
  LDH levels (UI/L) at the time of diagnosis will be compared
Comparison of splenomegaly proportion within the subtypes of clonal architecture | 24 months
  Proportion of patients with splenomegaly will be compared
Comparison of constitutional symptoms proportion within the subtypes of clonal architecture | 24 months
  Proportion of patients with constitutional symptoms will be compared
Evaluation of overall survival of the patients at 4 years according to their clonal architecture profile | 72 months
  Overall survival will be evaluated by Cox models
Evaluation of the leukemia-free survival of the patients at 4 years according to their clonal architecture profile | 72 months
  Leukemia-free survival will be evaluated by Cox models

CONTACTS AND LOCATIONS:
Overall Officials: POUILLART, Study Director — University Hospital, Angers
Locations (13):
- France (13):
  - CHU Angers, Angers
  - CHRU Brest, Brest
  - CH Cholet, Cholet
  - CHU Henri MONDOR, Créteil
  - Institut Paoli Calmettes, Marseille
  - CHU Nantes, Nantes
  - AP-HP Hôpital Saint Louis, Paris
  - Hôpital Bicêtre, Paris
  - CHU de Bordeaux, Pessac
  - CHU Lyon, Pierre-Bénite
  - CH de Cornouaille, Quimper
  - CHRU Tours - Hôpital Bretonneau, Tours
  - CH de Vannes, Vannes

IPD SHARING:
Plan to Share IPD: No